CLINICAL TRIAL: NCT03905694
Title: ILLUMINATE-B: An Open-Label Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Lumasiran in Infants and Young Children With Primary Hyperoxaluria Type 1
Brief Title: A Study of Lumasiran in Infants and Young Children With Primary Hyperoxaluria Type 1
Acronym: ILLUMINATE-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-GO1-004; 2018-004014-17 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Primary Hyperoxaluria; Primary Hyperoxaluria Type 1 (PH1)
Keywords: PH1; Primary Hyperoxaluria; Hyperoxaluria; RNAi Therapeutic; siRNA; AGT
MeSH Terms: conditions — Hyperoxaluria, Primary; Primary hyperoxaluria type 1; Hyperoxaluria | interventions — lumasiran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lumasiran (Experimental): Lumasiran will be administered by subcutaneous (SC) injection.
  Interventions: Drug: Lumasiran

INTERVENTIONS:
Drug: Lumasiran — Lumasiran will be administered by subcutaneous (SC) injection.
  Other Names: ALN-GO1

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of lumasiran in infants and young children with confirmed primary hyperoxaluria type 1 (PH1).

ELIGIBILITY:
Inclusion Criteria:

* Has genetic confirmation of primary hyperoxaluria type 1 (PH1)
* Meets urinary oxalate excretion requirements
* If taking Vitamin B6 (pyridoxine), must have been on stable regimen for at least 90 days

Exclusion Criteria:

* If <12 months old at screening, has an abnormally high serum creatinine
* If ≥12 months old at screening, has an estimated glomerular filtration rate (GFR) of ≤45 mL/min/1.73m^2
* Clinical evidence of systemic oxalosis
* History of kidney or liver transplant

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2024-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (9):
- United States (2):
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Houston, Texas
- France (2):
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Paris
- Clinical Trial Site, Bonn, Germany
- Israel (3):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Nahariya
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the United States (US) and/or the European Union (EU).
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Frishberg Y, Hayes W, Shasha-Lavsky H, Sas DJ, Michael M, Sellier-Leclerc AL, Hogan J, Willey R, Gansner JM, Magen D. Efficacy and safety of lumasiran for infants and young children with primary hyperoxaluria type 1: 30-month analysis of the phase 3 ILLUMINATE-B trial. Front Pediatr. 2024 Sep 16;12:1392644. doi: 10.3389/fped.2024.1392644. eCollection 2024. PMID 39355649
- [Derived] Hayes W, Sas DJ, Magen D, Shasha-Lavsky H, Michael M, Sellier-Leclerc AL, Hogan J, Ngo T, Sweetser MT, Gansner JM, McGregor TL, Frishberg Y. Efficacy and safety of lumasiran for infants and young children with primary hyperoxaluria type 1: 12-month analysis of the phase 3 ILLUMINATE-B trial. Pediatr Nephrol. 2023 Apr;38(4):1075-1086. doi: 10.1007/s00467-022-05684-1. Epub 2022 Aug 1. PMID 35913563
- [Derived] Sas DJ, Magen D, Hayes W, Shasha-Lavsky H, Michael M, Schulte I, Sellier-Leclerc AL, Lu J, Seddighzadeh A, Habtemariam B, McGregor TL, Fujita KP, Frishberg Y; ILLUMINATE-B Workgroup. Phase 3 trial of lumasiran for primary hyperoxaluria type 1: A new RNAi therapeutic in infants and young children. Genet Med. 2022 Mar;24(3):654-662. doi: 10.1016/j.gim.2021.10.024. Epub 2021 Dec 8. PMID 34906487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in France, Germany, Israel, the United Kingdom, and the United States from 22 April 2019 to 26 July 2024.
Pre-assignment Details: A total of 18 participants with Primary hyperoxaluria type 1 (PH1) were enrolled and treated in this study.
Groups:
- Lumasiran: Participants weighing <10 kg received loading doses of lumasiran subcutaneous (SC) injection 6.0 mg/kg monthly (QM) for 3 months, followed by maintenance doses of 3.0 mg/kg QM during the 6-month primary analysis period (PAP) & QM during the 54-month extension period (EP). Participants who transitioned from <10 kg to ≥10 kg continued monthly doses at 3.0 mg/kg until the next visit that coincided with a dose for participants weighing ≥10 kg. Thereafter, participants followed Q3M dosing until the end of the study.
  Participants weighing ≥10 to <20 kg received lumasiran 6.0 mg/kg QM for 3 months, then maintenance doses of 6.0 mg/kg at Months 3 & 6 in the 6-month PAP & Q3M during the 54-month EP.
  Participants ≥20 kg received lumasiran 3.0 mg/kg QM for 3 months, followed by maintenance doses of 3.0 mg/kg at Months 3 & 6 in the 6-month PAP & Q3M during the 54-month EP.
  Participants with weight increases to a new dosing category (<10 kg to ≥10 kg or <20 kg to ≥20 kg) followed the new regimen for the rest of the study or until the next dosing category threshold was reached; participants did not switch back to lower-weight dosing schedules if their body weight subsequently decreased.
Period: Primary Analysis Period
Arm/Group | Lumasiran
Started | 18
Completed | 18
Not Completed | 0
Period: Long-term Extension Period
Arm/Group | Lumasiran
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least one dose of Lumasiran during study.
Groups:
- Lumasiran: Participants weighing <10 kg received loading doses of lumasiran SC injection 6.0 mg/kg QM for 3 months, followed by maintenance doses of 3.0 mg/kg QM during the 6-month PAP & QM during the 54-month EP. Participants who transitioned from <10 kg to ≥10 kg continued monthly doses at 3.0 mg/kg until the next visit that coincided with a dose for participants weighing ≥10 kg. Thereafter, participants followed Q3M dosing until the end of the study.
  Participants weighing ≥10 to <20 kg received lumasiran 6.0 mg/kg QM for 3 months, then maintenance doses of 6.0 mg/kg at Months 3 & 6 in the 6-month PAP & Q3M during the 54-month EP.
  Participants ≥20 kg received lumasiran 3.0 mg/kg QM for 3 months, followed by maintenance doses of 3.0 mg/kg Months 3 & 6 in the 6-month PAP & Q3M during the 54-month EP.
  Participants with weight increases to a new dosing category (<10 kg to ≥10 kg or <20 kg to ≥20 kg) followed the new regimen for the rest of the study or until the next dosing category threshold was reached; participants did not switch back to lower-weight dosing schedules if their body weight subsequently decreased.
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: months] | 43.7 (21.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
Spot Urinary Oxalate:Creatinine Ratio [Mean (Standard Deviation); unit: mmol/mmol] | 0.6306 (0.42636)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Spot Urinary Oxalate:Creatinine Ratio From Baseline to Month 6
Description: Percent change in spot urinary oxalate:creatinine ratio was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: Efficacy Analysis Set: All participants who received any amount of lumasiran and had at least 1 valid spot urinary oxalate:creatinine ratio value at baseline and at least 1 valid spot urinary oxalate:creatinine ratio value from assessment(s) at Month 3 through Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percent change | -71.97 (2.706)
Statistical Analysis 1: Comparison: Lumasiran; Mixed-effect Model Repeated Measures (MMRM) includes scheduled visits (months 3, 4, 5, and 6) and baseline spot urinary oxalate:creatine ratio as fixed effects. Autoregressive (1) was used to model the within-patient error; Test type: Other — Not applied; Mixed model for repeated measures (MMRM); Least Squares (LS) Mean = -71.97, 95% CI 2-sided [-77.52 to -66.42]

2. Secondary Outcome: Percentage Change in Spot Urinary Oxalate: Creatinine Ratio in the Extension Period (Month 6 to End of Study [Month 60])
Description: A negative change from baseline indicates a favorable outcome.
Time Frame: From Month 6 to Month 60
Population: Efficacy analysis set included all participants who were treated with Lumasiran and had at least one spot urinary oxalate:creatinine ratio value at baseline and at least one spot urinary oxalate:creatinine ratio value from assessment(s) at Month 6 through Month 60.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percent change | -74.48 (4.246)

3. Secondary Outcome: Percentage of Time That Spot Urinary Oxalate: Creatinine Ratio is at or Below the Near-normalization Threshold (≤1.5 × Upper Limit of Normal (ULN) for Age)
Description: Percentage of time that spot urinary oxalate: creatinine (UOx:Cr) ratio level is at or below ≤ 1.5xULN is calculated as (cumulative months at or below near normalization threshold divided by cumulative months of assessments)*100. Cumulative months in near-normalization is defined as the summation across all intervals that met the near-normal threshold and cumulative months of valid assessments is defined as the summation across all valid post-baseline collections. ULN levels of spot urinary oxalate to creatinine ratio where urine oxalate levels were analyzed using enzymatic assay. The age-dependent reference ULN levels of spot urinary oxalate to creatinine ratio are as follows: 1-1.5 years=0.158; 1.5-2 years=0.138; 2-2.5 years=0.124; 2.5-3 years=0.116; 3-3.5 years=0.102; 3.5-4 years=0.094; 4-4.5 years=0.088; 4.5-5 years=0.082; 5-5.5 years=0.077; 5.5-6 years=0.073.
Time Frame: Up to 60 months
Population: Efficacy analysis set included all participants who were treated with Lumasiran and had at least one spot urinary oxalate:creatinine ratio value at baseline and at least one spot urinary oxalate:creatinine ratio value from assessment(s) throughout the study duration.
Measure: Median (Full Range); unit: percentage of time
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percentage of time | 68.95 [18.3 to 98.7]

4. Secondary Outcome: Absolute Change in Spot Urinary Oxalate: Creatinine Ratio From Baseline
Description: The absolute change is represented as ratio of millimoles of urinary oxalate to millimoles of urinary creatinine.
Time Frame: From Baseline to Month 6 and Month 60
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/mmol
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
mmol/mmol
  Month 6 | -0.4880 (0.09127)
  Month 60 | -0.5179 (0.09929)

5. Secondary Outcome: Percentage of Participants With Spot Urinary Oxalate: Creatinine Ratio Levels ≤ the ULN for Age
Description: The percentage of participants meeting the criteria (UOx:Cr ratio ≤ the ULN for age) at least at one post-baseline visit were reported for this outcome measure. The age-dependent reference ULN levels of spot urinary oxalate to creatinine ratio are as follows: 1-1.5 years=0.158; 1.5-2 years=0.138; 2-2.5 years=0.124; 2.5-3 years=0.116; 3-3.5 years=0.102; 3.5-4 years=0.094; 4-4.5 years=0.088; 4.5-5 years=0.082; 5-5.5 years=0.077; 5.5-6 years=0.073.
Time Frame: Up to 60 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percentage of participants | 100

6. Secondary Outcome: Percentage of Participants With Spot Urinary Oxalate: Creatinine Ratio Levels ≤ 1.5xULN for Age
Description: The percentage of participants meeting the criteria (UOx:Cr ratio ≤ 1.5xULN for age) at least at one post-baseline visit were reported for this outcome measure. The age-dependent reference ULN levels of spot urinary oxalate to creatinine ratio are as follows: 1-1.5 years=0.158; 1.5-2 years=0.138; 2-2.5 years=0.124; 2.5-3 years=0.116; 3-3.5 years=0.102; 3.5-4 years=0.094; 4-4.5 years=0.088; 4.5-5 years=0.082; 5-5.5 years=0.077; 5.5-6 years=0.073.
Time Frame: Up to 60 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percentage of participants | 100

7. Secondary Outcome: Percentage Change in Plasma Oxalate From Baseline to End of Study (Month 60)
Description: The lower limit of quantification (LLOQ) was 5.55 micromoles per liter (μmol/L). A negative change from baseline indicates a favorable outcome.
Time Frame: From Baseline to Month 6 and Month 60
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
percent change
  Month 6 | -32.06 (6.711)
  Month 60 | -24.78 (12.814)

8. Secondary Outcome: Absolute Change in Plasma Oxalate From Baseline to End of Study (Month 60)
Description: The LLOQ was 5.55 μmol/L. A negative change from Baseline indicates a favorable outcome.
Time Frame: From Baseline to Month 6 and Month 60
Population: as for outcome 3
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
µmol/L
  Month 6 | -5.03 (1.294)
  Month 60 | -5.03 (1.859)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lumasiran
Description: Cmax was the maximum plasma concentration post-dose within the pharmacokinetic (PK) sampling time frame. Higher Cmax generally indicates higher drug exposure.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: PK analysis set included all participants who had received at least one full dose of Lumasiran and had at least one post-dose blood sample for PK parameters and had evaluable PK data. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
nanograms per milliliter (ng/mL)
  Day 1 | 886 (58.9)
  Month 6 | 869 (84.0)
  Month 12: number analyzed (Participants) | 17
  Month 12 | 1180 (83.5)
  Month 18 | 878 (94.0)
  Month 24: number analyzed (Participants) | 17
  Month 24 | 790 (91.9)

10. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Lumasiran
Description: Tmax was estimated by calculating the time required to reach the maximum plasma concentration (Cmax) after the drug administration. Lower Tmax generally indicates faster drug absorption from the administration site.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 9
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
hours (h)
  Day 1 | 3.74 [1.87 to 8.1]
  Month 6 | 4 [1.75 to 10.1]
  Month 12: number analyzed (Participants) | 17
  Month 12 | 4 [1.75 to 7.25]
  Month 18 | 3.64 [1.98 to 10]
  Month 24: number analyzed (Participants) | 17
  Month 24 | 3.73 [1.67 to 10.3]

11. Secondary Outcome: Elimination Half-life (t1/2beta) of Lumasiran
Description: Elimination half-life was estimated from the terminal phase of the plasma concentration-time profile post-dose. Shorter half-life generally indicates rapid drug elimination from the body.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: PK analysis set included all participants who had received at least one full dose of Lumasiran and had at least one post-dose blood sample for PK parameters and had evaluable PK data. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Lumasiran
Number analyzed (Participants) | 13
hours (h)
  Day 1 | 5.46 [1.42 to 10.3]
  Month 6: number analyzed (Participants) | 8
  Month 6 | 5.96 [3.04 to 9]
  Month 12: number analyzed (Participants) | 8
  Month 12 | 3.52 [1.56 to 6.64]
  Month 18: number analyzed (Participants) | 9
  Month 18 | 3.74 [1.62 to 13.9]
  Month 24: number analyzed (Participants) | 8
  Month 24 | 4.99 [2.69 to 10.8]

12. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours (AUC0-24) of Lumasiran
Description: AUC0-24 was the total drug exposure calculated as the area under the plasma concentration-time curve from the time of dosing (t = 0) to 24 hours.
Time Frame: 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Lumasiran
Number analyzed (Participants) | 14
hours*nanograms per milliliter (h*ng/mL)
  Day 1 | 8050 (37.7)
  Month 6: number analyzed (Participants) | 11
  Month 6 | 8450 (41.1)
  Month 12: number analyzed (Participants) | 12
  Month 12 | 10800 (39.3)
  Month 18: number analyzed (Participants) | 12
  Month 18 | 8420 (57.2)
  Month 24 | 7420 (61.6)

13. Secondary Outcome: Area Under the Concentration-time Curve From 0 to Last Quantifiable Concentration (AUC0-last) of Lumasiran
Description: AUC0-last was the total drug exposure calculated as the area under the plasma concentration-time curve from time 0 to the time of the last measurable (quantifiable) concentration (C_last).
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
h*ng/mL
  Day 1 | 7870 (33.4)
  Month 6 | 6620 (95.5)
  Month 12: number analyzed (Participants) | 17
  Month 12 | 8480 (76.1)
  Month 18 | 5770 (155.0)
  Month 24: number analyzed (Participants) | 17
  Month 24 | 7100 (80.0)

14. Secondary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC0-infinity) of Lumasiran
Description: AUC0-infinity was the total drug exposure estimated as the area under the plasma concentration-time curve from time 0 extrapolated to infinity.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lumasiran
Number analyzed (Participants) | 13
h*ng/mL
  Day 1 | 9180 (31.7)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 8840 (40.9)
  Month 12: number analyzed (Participants) | 8
  Month 12 | 11900 (29.2)
  Month 18: number analyzed (Participants) | 9
  Month 18 | 11600 (48.6)
  Month 24: number analyzed (Participants) | 8
  Month 24 | 9610 (48.8)

15. Secondary Outcome: Apparent Clearance (CL/F) of Lumasiran
Description: Apparent clearance was calculated by dividing the area under the plasma concentration-time curve from zero infinity by the dose administered. A higher clearance generally indicates faster elimination from the body.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Lumasiran
Number analyzed (Participants) | 13
liters per hour (L/h)
  Day 1 | 8.62 (24.0)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 10.2 (32.3)
  Month 12: number analyzed (Participants) | 8
  Month 12 | 7.06 (28.3)
  Month 18: number analyzed (Participants) | 9
  Month 18 | 6.87 (30.6)
  Month 24: number analyzed (Participants) | 8
  Month 24 | 8.22 (37.7)

16. Secondary Outcome: Apparent Volume of Distribution (V/F) of Lumasiran
Description: Apparent Volume of Distribution generally indicates the extent of drug distribution in the body.
Time Frame: 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose on Day 1, Month 6, Month 12, Month 18 and Month 24
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Lumasiran
Number analyzed (Participants) | 13
Liters (L)
  Day 1 | 57.2 (69.8)
  Month 6: number analyzed (Participants) | 8
  Month 6 | 81 (71.1)
  Month 12: number analyzed (Participants) | 8
  Month 12 | 36 (75.6)
  Month 18: number analyzed (Participants) | 9
  Month 18 | 43.1 (107.1)
  Month 24: number analyzed (Participants) | 8
  Month 24 | 57.6 (70.6)

17. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR [in milliliters per minute per 1.73 meters square (mL/min/1.73m^2)] was calculated from serum creatinine (SCr) based on the Schwartz Bedside Formula for participants ≥12 months of age at the time of assessment.
Time Frame: From Baseline to Month 6 and Month 60
Population: Efficacy analysis set included all participants who were treated with Lumasiran and had at least one spot urinary oxalate:creatinine ratio value at baseline and at least one spot urinary oxalate:creatinine ratio value from assessment(s) throughout the study duration. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Lumasiran
Number analyzed (Participants) | 16
mL/min/1.73m^2
  Month 6 | -0.263 (3.8461)
  Month 60 | -4.525 (4.8873)

18. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 60 months
Population: Safety analysis set included all participants who had received at least one dose of Lumasiran.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumasiran
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to 60 months
Description: Safety analysis set included all subjects who had received at least one dose of Lumasiran.
Arm/Group | Lumasiran
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumasiran (N=18)
Viral infection (Infections and infestations) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumasiran (N=18)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Microcytosis (Blood and lymphatic system disorders) | 1 (1)
Factor XII deficiency (Congenital, familial and genetic disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 4 (5)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anal pruritus (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Dental caries (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Teething (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (13)
Fatigue (General disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (3)
Injection site haematoma (General disorders) | 1 (2)
Injection site reaction (General disorders) | 3 (4)
Injection site urticaria (General disorders) | 1 (2)
Pyrexia (General disorders) | 8 (16)
Vessel puncture site haematoma (General disorders) | 1 (2)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3)
COVID-19 (Infections and infestations) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 3 (4)
Eye infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 4 (5)
Nasopharyngitis (Infections and infestations) | 4 (14)
Oral herpes (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 2 (4)
Pharyngitis (Infections and infestations) | 3 (4)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 5 (10)
Streptococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (9)
Urinary tract infection (Infections and infestations) | 3 (3)
Varicella (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3)
SARS-CoV-2 antibody test positive (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Behaviour disorder (Psychiatric disorders) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Blood creatinine increased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is intended that after completion of the study, the data are to be submitted for publication in a scientific journal and/or for reporting at a scientific meeting. A separate publication by Institution or PI may not be submitted for publication until after this primary manuscript is published or following 12 months after completion of the study. A copy of any proposed publication based on this study, must be provided and confirmed received at the Sponsor at least 30 days before its submission.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03905694/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT03905694/SAP_002.pdf